CLINICAL TRIAL: NCT07198737
Title: Effect of Virtual Reality and Trans Auricular X-Vagus Nerve Stimulation for Anxiety and Depression in Chronic Shoulder Pain Patients
Acronym: VIRTAX-ADSP
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: East Kent Hospitals University NHS Foundation Trust (Other Government)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Device Feasibility
Other Study IDs: S2024-CTU14-MH
Record Dates: First submitted 2025-09-22; First posted 2025-09-30 (Actual); Last update posted 2025-09-30 (Actual); Status verified 2025-09

CONDITIONS: Chronic Pain (Back / Neck)
Keywords: VR VNS
MeSH Terms: conditions — Chronic Pain

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Treatment with VR/VNS (Experimental)
  Interventions: Device: VR and VNS

INTERVENTIONS:
Device: VR and VNS — Participants will have Vagus nerve stimulation at the same time as a relaxing VR experience

SUMMARY:
Chronic shoulder pain is a debilitating condition that significantly impacts quality of life, daily functioning, and mental well-being. For individuals awaiting surgical intervention for a long period, prolonged pain often leads to heightened psychological distress, poor sleep quality, and reduced overall health outcomes. Innovative approaches are urgently needed to address these challenges and improve preoperative management.

This study will combine 2 technologies which have both been shown to help relax and calm users.

Transcutaneous Auricular Vagus Nerve Stimulation (taVNS) is

* a gentle non-invasive therapy that uses a small device to send tiny electrical pulses to a spot on your outer ear. The principle of using electrical pulses are similar to pacemaker or TENS machines.
* These pulses help stimulate a special nerve called the vagus nerve, which is like a superhighway between your brain and your body

Your vagus nerve helps control:

* Your mood and anxiety levels
* Healing of nerves and other organs in the body
* How your body handles pain
* Digestion, heart rate, and more By stimulating the vagus nerve, taVNS can help your body relax, reset, and feel better.

While virtual reality (VR) has demonstrated effectiveness in distracting from pain and improving psychological resilience.

These two will be combined so that the participant experiences a relaxing VR environment that helps them control their breathing while receiving taVNS. With the aim of managing chronic pain by targeting both physical and psychological dimensions.

This study aims to evaluate the feasibility and safety, of a trial of taVNS paired with VR looking at trial recruitment, retention and compliance. Secondary to this the study will look to see if there is evidence of taVNS +VR in reducing pain, enhancing psychological well-being, and improving quality of life for individuals with chronic shoulder pain awaiting surgery. It will provide critical insights into the potential of this combined intervention as a preoperative and potentially post operative pain management strategy.

ELIGIBILITY:
Inclusion Criteria:

* Aged over 18.
* Ability to understand English
* Ability to provide informed consent and attend in-person sessions
* Chronic shoulder pain (pain lasting for at least 6 months) waiting on surgical pathway.
* Comorbid mild-to-moderate anxiety or depression
* Referred by a consultant orthopaedic surgeon.
* Unresponsive to conventional treatment for 6 months including antidepressants, physiotherapy, and/ or oral analgesics
* Mean NRS pain score ≥ 5 on most or all days either continuously or in motion

Exclusion Criteria:● Inability to understand English and consent process

* History of significant neurological or psychiatric conditions unrelated to chronic pain (e.g., epilepsy, psychosis, schizophrenia).
* Skin lesions or piercing or extensive tattooing of the concha or Skin disease: infection, eczema or cancer of the ears or skin in region where VR headset or taVNS would sit
* Presence of active implants (e.g. cochlear implant, implanted vagus nerve stimulator, cardiac pacemaker, implantable cardioverter defibrillator (ICD) deep brain stimulations or spinal cord stimulators, ventriculoperitoneal (VP) shunt).
* Inability to tolerate VR (e.g., severe motion sickness, vertigo or balance issues, claustrophobia).
* Fear of heights
* Active infections, significant trauma, or other acute conditions affecting the shoulder.
* Pregnancy and women trying actively to conceive
* Pre-existing Persistent post-surgical pain-(>6 months) from surgeries other than shoulder replacements
* On- going alcohol and/ or drug problem
* Widespread chronic pain conditions (fibromyalgia, complex regional pain syndrome)
* Involvement in any clinical studies within the last 28 days prior to assessment
* Other therapies such as other psychological interventions for A/D and pain in the shoulder are not allowed for the period of the study and follow up unless there is a psychiatric emergency. Participants may also not be involved in any trial on pain management or related to shoulders while participating in this VR/VNS trial.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Estimated)
Dates: Start 2025-11-01 (Estimated); Primary Completion 2026-07-01 (Estimated); Study Completion 2026-08-01 (Estimated)

PRIMARY OUTCOMES:
Recruitment and retention rates | from enrolment to the end of treatment at 5 weeks
  The proportion of eligible participants successfully enrolled in eth study and the percentage who remain in the study until its conclusion

CONTACTS AND LOCATIONS:
Locations (1):
- East kent Clinical trials Unit, Margate, Kent, United Kingdom

IPD SHARING:
Plan to Share IPD: No